CLINICAL TRIAL: NCT00641069
Title: Effect on Hemodynamics of Automated Band Chest Compression Device in Cardiac Arrest Resuscitation
Brief Title: Automated Chest Compression in Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Beaujon Hospital (Other)
Responsible Party: François-Xavier Duchateau, MD, Departement of Anesthesiology, Intensive Care and EMS, Beaujon Hospital
Other Study IDs: BAND V6
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Automated load-distributing band device — Blood pressure recording before and after starting up the automated band device
  Other Names: AutoPulse™ 100, Zoll®

SUMMARY:
To evaluate the effect of use of automated chest compression device on blood pressure in patients presenting with cardiac arrest. Higher systolic, diastolic and mean blood pressures are expected.

DETAILED DESCRIPTION:
The protocol compares arterial pressures produced by an automated self-adjusting load-distributing band device (AutoPulse™ 100, Zoll®) with those of manual cardiopulmonary resuscitation in refractory out-of-hospital cardiac arrest. Each patient will receive first manual compressions and then automated resuscitation.

Patients presenting with cardiac arrest are treated following standard advanced life support guidelines. They are intubated and ventilated, received epinephrine and defibrillation if appropriate. Manuel chest compressions are continued. An arterial catheter is placed to monitor hemodynamics continuously as we usually do in this case. Patients are included at this stage. Three blood pressure values (every 1 minutes) are recorded. Then, the automated band device is started up without any pause, following our procedure for refractory cardiac arrest. Three blood pressure values are recorded again, during automated cardiopulmonary resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Refractory cardiac arrest

Exclusion Criteria:

* Defective invasive arterial blood pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18 with out-of-hospital cardiac arrest
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Diastolic blood pressures produced by manual and then by automated chest compressions will be recorded for each patient | Instantaneously

SECONDARY OUTCOMES:
Systolic blood pressures produced by manual and then by automated chest compressions will be recorded for each patient | Instantaneously
Mean blood pressures produced by manual and then by automated chest compressions will be recorded for each patient | Instantaneously

CONTACTS AND LOCATIONS:
Overall Officials: Francois-Xavier Duchateau, MD, Principal Investigator — Departement of Anesthesiology, Intensive Care and EMS, Beaujon University Hospital; Jean Mantz, MDPhD, Study Chair — Departement of Anesthesiology, Intensive Care and EMS, Beaujon University Hospital
Locations (1):
- Departement of Anesthesiology, Intensive Care and EMS, Beaujon University Hospital, Clichy, France